CLINICAL TRIAL: NCT02573324
Title: A Randomized, Placebo Controlled Phase 3 Study of ABT-414 With Concurrent Chemoradiation and Adjuvant Temozolomide in Subjects With Newly Diagnosed Glioblastoma (GBM) With Epidermal Growth Factor Receptor (EGFR) Amplification (Intellance1)
Brief Title: A Study of ABT-414 in Participants With Newly Diagnosed Glioblastoma (GBM) With Epidermal Growth Factor Receptor (EGFR) Amplification
Acronym: Intellance1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M13-813; 2015-001166-26 (EudraCT Number)
Expanded Access: NCT03123952 (No longer available)
Record Dates: First submitted 2015-09-28; First posted 2015-10-09 (Estimated); Results first posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Newly Diagnosed Glioblastoma; Epithelial Growth Factor Receptor (EGFR); Temozolomide; ABT-414; Radiology Therapy Oncology Group; Antibody Drug Conjugate; Brain Tumor; Brain Tumor Group; EGFRvIII; EGFR Amplified; First Line Therapy; Brain Cancer
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Temozolomide; depatuxizumab mafodotin; ABT-414; Radiation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sub-study was open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Depatuxizumab Mafodotin, Radiation and Temozolomide (TMZ) (Experimental): Depatuxizumab mafodotin is given on Day 1 of Week 1, 3 and 5 along with the standard therapy of TMZ and radiation during the chemoradiation phase. Depatuxizumab mafodotin is given on Day 1 and 15 of each cycle along with TMZ (Days 1-5 of each cycle) per standard of care during the adjuvant phase.
  Interventions: Drug: Temozolomide; Drug: Depatuxizumab mafodotin; Radiation: Radiation
- Placebo, Radiation and TMZ (Placebo Comparator): Placebo is given on Day 1 of Week 1, 3 and 5 along with the standard therapy of TMZ and radiation during the chemoradiation phase. Placebo is given on Day 1 and 15 of each cycle along with TMZ (Days 1-5 of each cycle) per standard of care during the adjuvant phase.
  Interventions: Drug: Temozolomide; Radiation: Radiation; Drug: Placebo for ABT-414
- Open-Label Sub-Study: Depatuxizumab Mafodotin, Radiation and TMZ (Experimental): Depatuxizumab mafodotin is given to participants with hepatic impairment on Day 1 of Week 1, 3 and 5 along with the standard therapy of TMZ and radiation during the chemoradiation phase. Depatuxizumab mafodotin is given on Day 1 and 15 of each cycle along with TMZ (Days 1-5 of each cycle) per standard of care during the adjuvant phase.
  Interventions: Drug: Temozolomide; Drug: Depatuxizumab mafodotin; Radiation: Radiation

INTERVENTIONS:
Drug: Temozolomide — Oral Capsule
Drug: Depatuxizumab mafodotin — Intravenous (IV) Infusion
  Other Names: ABT-414
  Arms: Depatuxizumab Mafodotin, Radiation and Temozolomide (TMZ); Open-Label Sub-Study: Depatuxizumab Mafodotin, Radiation and TMZ
Radiation: Radiation
Drug: Placebo for ABT-414 — IV Infusion (IV)
  Arms: Placebo, Radiation and TMZ

SUMMARY:
This study seeks to determine whether the addition of ABT-414 to concomitant radiotherapy and temozolomide (TMZ) followed by combination of ABT-414 with adjuvant TMZ prolongs overall survival (OS) among participants with newly diagnosed glioblastoma (GBM) with epidermal growth factor receptor (EGFR) amplification.

In addition, there is a Phase 1, open-label, multicenter sub-study to assess the pharmacokinetics, safety and tolerability of ABT-414 in participants with newly diagnosed EGFR-amplified GBM who have mild or moderate hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical diagnosis of glioblastoma (GBM).
* Must have a confirmed epidermal growth factor receptor amplification in tumor tissue.
* Must have a Karnofsky Performance Status (KPS) >= 70 at assessment <= 14 days prior to randomization (N/A to the sub-study).
* Must have recovered from effects of surgery, postoperative infection and other complications of surgery.
* Must have adequate bone marrow, renal, and hepatic function (For the sub-study, the participant must have adequate bone marrow and renal function and have mild-to-moderate hepatic impairment).

Exclusion Criteria:

* Multifocal, recurrent or metastatic GBM or gliomatosis cerebri (For the sub-study, the participant can have multifocal GBM and glimatosis cerebri but can't have recurrent or metastatic GBM).
* Prior chemo therapy or radiosensitizer for head and neck cancer.
* Prior radiotherapy to the head or neck in overlap of radiation fields.
* Prior therapy for glioblastoma or other invasive malignancy.
* Prior, concomitant or planned treatment with Novo Tumor Treatment Fields (Novo-TTF), EGFR-targeted therapy, bevacizumab, Gliadel wafers or other intratumoral or intracavity anti-neoplastic therapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 691 (Actual)
Dates: Start 2015-01-04 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (212):
- United States (68):
  - St. Josephs Hospital and Med Center /ID# 144149, Phoenix, Arizona
  - Highlands Oncology Group, PA /ID# 142050, Springdale, Arkansas
  - University of Southern California /ID# 147543, Los Angeles, California
  - University of California, Los Angeles /ID# 149239, Los Angeles, California
  - Sharp Memorial Hospital /ID# 148193, San Diego, California
  - Univ California, San Francisco /ID# 145889, San Francisco, California
  - Duplicate_St. John's Health Center /ID# 148192, Santa Monica, California
  - Cedars-Sinai Medical Center-West Hollywood /ID# 148472, West Hollywood, California
  - Univ of Colorado Cancer Center /ID# 148194, Aurora, Colorado
  - Associated Neurologists of Sou /ID# 147701, Fairfield, Connecticut
  - Yale University /ID# 144170, New Haven, Connecticut
  - Christiana Care Health Service /ID# 144127, Newark, Delaware
  - Boca Raton Regional Hospital /ID# 163659, Boca Raton, Florida
  - Holy Cross Hospital /ID# 156764, Fort Lauderdale, Florida
  - Baptist Hospital Miami /ID# 152451, Miami, Florida
  - Advent Health /ID# 144128, Orlando, Florida
  - Moffitt Cancer Center /ID# 144130, Tampa, Florida
  - Piedmont Hospital /ID# 145892, Atlanta, Georgia
  - Emory Midtown Infectious Disease Clinic /ID# 144015, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 147895, Chicago, Illinois
  - The University of Chicago Medical Center /ID# 144158, Chicago, Illinois
  - NorthShore University HealthSystem /ID# 144017, Evanston, Illinois
  - Northwestern Medicine Cancer Center - Warrenville /ID# 148476, Warrenville, Illinois
  - Parkview Research Ctr, Hosp /ID# 144150, Fort Wayne, Indiana
  - Univ Kansas Cancer Ctr - Overl /ID# 145895, Westwood, Kansas
  - Maine Medical Partners Neurolo /ID# 160864, Scarborough, Maine
  - Tufts Medical Center /ID# 145897, Boston, Massachusetts
  - Massachusetts General Hospital /ID# 144145, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 148475, Boston, Massachusetts
  - Wayne State University /ID# 145890, Detroit, Michigan
  - Henry Ford Health System /ID# 145896, Detroit, Michigan
  - Duplicate_St. Joseph Mercy Hospital /ID# 144143, Ypsilanti, Michigan
  - Mmcorc /Id# 144146, Saint Louis Park, Minnesota
  - Washington University-School of Medicine /ID# 144174, St Louis, Missouri
  - Nebraska Methodist Hospital /ID# 144140, Omaha, Nebraska
  - University of Nebraska Medical Center /ID# 145899, Omaha, Nebraska
  - MD Anderson Cancer Center at Cooper - Camden /ID# 145891, Camden, New Jersey
  - Rutgers Cancer Institute of New Jersey /ID# 148190, New Brunswick, New Jersey
  - Columbia University Medical Center /ID# 144020, New York, New York
  - University of Rochester Medical Center /ID# 144166, Rochester, New York
  - Levine Cancer Ins, Carolina Me /ID# 144124, Charlotte, North Carolina
  - University of Cincinnati /ID# 144164, Cincinnati, Ohio
  - Duplicate_Univ Hosp Cleveland /ID# 144153, Cleveland, Ohio
  - Cleveland Clinic Main Campus /ID# 144023, Cleveland, Ohio
  - The Ohio State University /ID# 144016, Columbus, Ohio
  - University of Toledo /ID# 156763, Toledo, Ohio
  - Univ Oklahoma HSC /ID# 144161, Oklahoma City, Oklahoma
  - St. Luke's Hospital /ID# 148191, Bethlehem, Pennsylvania
  - Penn State University and Milton S. Hershey Medical Center /ID# 147525, Hershey, Pennsylvania
  - University of Pennsylvania /ID# 157623, Philadelphia, Pennsylvania
  - Thomas Jefferson University /ID# 144191, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center /ID# 145893, Philadelphia, Pennsylvania
  - Allegheny General Hospital /ID# 144126, Pittsburgh, Pennsylvania
  - University of Pennsylvania Medical Center - Shadyside /ID# 144159, Pittsburgh, Pennsylvania
  - Medical University of South Carolina /ID# 144141, Charleston, South Carolina
  - Austin Cancer Centers /ID# 151061, Austin, Texas
  - Baylor Sammons Cancer Center /ID# 155542, Dallas, Texas
  - The University of Texas Health Science Center at Houston /ID# 144013, Houston, Texas
  - University of Texas MD Anderson Cancer Center /ID# 144018, Houston, Texas
  - Duplicate_Scott and White Medical Center /ID# 160743, Temple, Texas
  - Intermountain Medical Center /ID# 144142, Murray, Utah
  - University of Utah /ID# 144160, Salt Lake City, Utah
  - Inova Health System /ID# 152956, Falls Church, Virginia
  - Virginia Commonwealth University Medical Center Main Hospital /ID# 149014, Richmond, Virginia
  - Virginia Mason Medical Center /ID# 144022, Seattle, Washington
  - University of Washington /ID# 144162, Seattle, Washington
  - Univ of Wisconsin Hosp/Clinics /ID# 144167, Madison, Wisconsin
  - Froedtert Memorial Lutheran Hospital /ID# 144139, Milwaukee, Wisconsin
- Argentina (2):
  - Sanatorio Parque /ID# 142825, Rosario, Santa Fe Province
  - Duplicate_Instituto Med Alex Flem /ID# 142884, Buenos Aires
- Australia (11):
  - Liverpool Hospital /ID# 144392, Liverpool, New South Wales
  - Duplicate_The Prince of Wales Hospital /ID# 144882, Randwick, New South Wales
  - Royal North Shore Hospital /ID# 143870, St Leonards, New South Wales
  - Calvary Mater Newcastle /ID# 143860, Waratah, New South Wales
  - Southern Medical Day Care Centre /ID# 143868, Wollongong, New South Wales
  - Princess Alexandra Hospital /ID# 143857, Woolloongabba, Queensland
  - Royal Adelaide Hospital /ID# 143867, Adelaide, South Australia
  - Calvary North Adelaide Hospita /ID# 143866, Adelaide, South Australia
  - St Vincent's Hospital Melbourne /ID# 143858, Fitzroy Melbourne, Victoria
  - Duplicate_Austin Hospital /ID# 143859, Heidelberg, Victoria
  - St John Of God Subiaco Hospital /ID# 143869, Subiaco, Western Australia
- Austria (4):
  - Medizinische Universitaet Graz /ID# 141982, Graz, Styria
  - Medizinische Universitaet Wien /ID# 141981, Vienna, Vienna
  - Duplicate_Medizinische Universitat Innsbruck,Universitatsklinik fur Innere Mediz /ID# 141984, Innsbruck
  - Kepler Universitätsklinikum GmbH - Neuromed Campus /ID# 141983, Linz
- Belgium (7):
  - UCL Saint-Luc /ID# 141648, Woluwe-Saint-Lambert, Brussels Capital
  - Grand Hopital de Charleroi /ID# 141645, Charleroi, Hainaut
  - UZ Gent /ID# 141647, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 143872, Leuven, Vlaams-Brabant
  - Duplicate_Centre Hospitalier Jolimont /ID# 143873, La Louvière
  - CHU de Liege /ID# 162860, Liège
  - Duplicate_UCL Mont Godinne /ID# 141644, Yvoir
- Brazil (5):
  - Liga Norte Riograndense Contra o Câncer /ID# 143878, Natal, Rio Grande do Norte
  - Hospital Sao Lucas da PUCRS /ID# 143879, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos /ID# 143876, Barretos, São Paulo
  - Instituto do Câncer do Estado de São Paulo - ICESP /ID# 144031, São Paulo, São Paulo
  - Instituto Nacional de Câncer José Alencar Gomes da Silva (INCA) /ID# 143877, Rio de Janeiro
- Canada (12):
  - Duplicate_Cancer Care Manitoba /ID# 149253, Winnipeg, Manitoba
  - QE II Health Sciences Centre /ID# 151600, Halifax, Nova Scotia
  - Juravinski Cancer Centre /ID# 152117, Hamilton, Ontario
  - Victoria Hospital /ID# 144184, London, Ontario
  - Ottawa Hospital Research Institute /ID# 150120, Ottawa, Ontario
  - Princess Margaret Cancer Centre /ID# 166277, Toronto, Ontario
  - Duplicate_Hospital Maisonneuve-Rosemont /ID# 149315, Montreal, Quebec
  - CHUM - Notre-Dame Hospital /ID# 144027, Montreal, Quebec
  - Duplicate_Jewish General Hospital /ID# 144029, Montreal, Quebec
  - Royal Victoria Hospital / McGill University Health Centre /ID# 144187, Montreal, Quebec
  - CHU de Quebec-Universite Laval /ID# 144189, Québec, Quebec
  - CHUS - Hopital Fleurimont /ID# 149771, Sherbrooke, Quebec
- China (14):
  - Anhui Provincial Hospital /ID# 166320, Hefei, Anhui
  - SanboBrain Hospital Capital Medical University /ID# 166422, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital /ID# 157430, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Center /ID# 143919, Guangzhou, Guangdong
  - Tongji Hospital Tongji Medical College of HUST /ID# 163820, Wuhan, Hubei
  - Duplicate_Xiangya Hospital Central South University /ID# 166791, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University /ID# 165596, Suzhou, Jiangsu
  - Duplicate_Tangdu Hospital /ID# 143920, Xi'an, Shaanxi
  - Duplicate_Huashan Hospital of Fudan University /ID# 159999, Shanghai, Shanghai Municipality
  - Duplicate_The Second Affiliated Hospital of ZUSM /ID# 165593, Hangzhou, Zhejiang
  - Beijing Tian Tan Hospital, Capital Medical University /ID# 167160, Beijing
  - The First Affiliated Hospital of Fujian Medical University /ID# 159166, Fuzhou
  - Duplicate_Shengjing Hospital of China Medical University /ID# 167016, Shenyang
  - Duplicate_Tianjin Med Univ General Hosp /ID# 143923, Tianjin
- Colombia (5):
  - Hospital Pablo Tobon Uribe /ID# 143780, Medellín, Antioquia
  - Administradora del Country_S.A-Clinica Del Country /ID# 143881, Bogota, Cundinamarca
  - Instituto Medico de Alta Tecnologia Oncomédica S.A /ID# 147223, Montería, Departamento de Córdoba
  - Oncologos del Occidente S.A /ID# 147713, Pereira, Risaralda Department
  - Centro Medico Imbanaco de Cali /ID# 143882, Cali
- Czechia (5):
  - Masarykuv onkologicky ustav /ID# 143884, Brno
  - Duplicate_FN Hradec Kralove /ID# 143885, Hradec Králové
  - Krajska nemocnice Liberec, a.s. /ID# 142024, Liberec
  - Duplicate_Univ Hosp Ostrava-Poruba /ID# 143883, Ostrava
  - Fakultni Nemocnice v Motole /ID# 142023, Prague
- France (8):
  - AP-HM - Hopital de la Timone /ID# 143911, Marseille, Bouches-du-Rhone
  - CHRU Lille - Hopital Claude Huriez /ID# 143915, Lille, Hauts-de-France
  - Institut de Cancérologie de l'Ouest René Gauducheau /ID# 143914, Saint-Herblain, Loire-Atlantique
  - CHU Nice -Hopital Pasteur /ID# 143916, Nice, Provence-Alpes-Côte d'Azur Region
  - Insititut de Cancerologie /ID# 143908, Angers
  - Hopital Pitie Salpetriere /ID# 143917, Paris
  - Hopital Avicenne - APHP /ID# 143910, Bobigny, Île-de-France Region
  - Duplicate_Gustave Roussy /ID# 143912, Villejuif, Île-de-France Region
- Germany (4):
  - Universitaetsklinik Heidelberg /ID# 143927, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 143926, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Leipzig /ID# 143962, Leipzig, Saxony
  - Universitaetsklinikum Knappschaftskrankenhaus Bochum GmbH /ID# 143961, Bochum
- Prince of Wales Hospital /ID# 143952, Hong Kong, Hong Kong
- Beaumont Hospital /ID# 142969, Beaumont, Dublin, Ireland
- Israel (5):
  - The Chaim Sheba Medical Center /ID# 143960, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 143956, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 143959, Haifa
  - Gastroenterology Institute, Division of Medicine /ID# 143958, Jerusalem
  - Rabin Medical Center /ID# 143957, Petah Tikva
- Italy (4):
  - Duplicate_Duplicate_AOU Citta della Salute Scienza /ID# 141801, Turin, Piedmont
  - Fondazione IRCCS Istituto Neurologico Carlo Besta /ID# 141800, Milan
  - Istituto Oncologico Veneto /ID# 143821, Padua
  - Duplicate_Regina Elena National Cancer I /ID# 141795, Rome
- Centro Medico Zambrano Hellion /ID# 143845, San Pedro Garza García, Nuevo León, Mexico
- Netherlands (5):
  - Vrije Universiteit Medisch Centrum /ID# 143889, Amsterdam
  - Universitair Medisch Centrum Groningen /ID# 141408, Groningen
  - Maastricht Universitair Medisch Centrum /ID# 143585, Maastricht
  - Haaglanden Medisch Centrum /ID# 141405, The Hague
  - Universitair Medisch Centrum Utrecht /ID# 141406, Utrecht
- New Zealand (2):
  - Duplicate_Canterbury District Health Boa /ID# 143861, Christchurch
  - Duplicate_Wellington Hospital (Capital and Coast District Health Board) /ID# 143890, Wellington
- Portugal (5):
  - CCA Braga - Hospital de Braga /ID# 141940, Braga
  - Centro Hospitalar Universitário do Algarve, EPE - Hospital Faro /ID# 141939, Faro
  - IPO Lisboa FG, EPE /ID# 141938, Lisbon
  - Centro Hospitalar Universitario de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 141941, Lisbon
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 142830, Porto
- Russia (7):
  - Regional Clinical Hospital of Kaliningrad region /ID# 141702, Kaliningrad, Kaliningrad Oblast
  - State budgetary healthcare institution Republican Clinical Oncology Dispensary /ID# 141706, Ufa, Kirov Oblast
  - Federal State Budgetary Scientific Institution N.N. Blokhin /ID# 141707, Moscow, Moscow
  - National Medical Research Center for Neurosurgery n.a. N. N. Burdenko /ID# 141701, Moscow, Moscow
  - Federal State Treatment and Rehabilitation center /ID# 141704, Moscow, Moscow
  - GEMC - European Medical Center /ID# 141703, Moscow, Moscow Oblast
  - Sverdlovsk Regional Oncology Dispensary /ID# 141700, Yekaterinburg, Sverdlovsk Oblast
- Singapore (2):
  - National University Hospital /ID# 143933, Singapore
  - National Cancer Ctr Singapore /ID# 143932, Singapore
- South Africa (6):
  - University of Free State, Universitas Annex (National Hospital Grounds) /ID# 144064, Bloemfontein, Free State
  - Netcare Unitas Hospital /ID# 152936, Centurion, Gauteng
  - The Oncology Centre /ID# 143950, Durban, KwaZulu-Natal
  - Netcare Oncology Intervent Ctr /ID# 143951, Cape Town, Western Cape
  - Rondebosch Oncology Center /ID# 143949, Cape Town, Western Cape
  - Cape Town Oncology Trials /ID# 143948, Kraaifontein, Western Cape
- South Korea (5):
  - National Cancer Center /ID# 141845, Goyang, Gyeonggido
  - Duplicate_Yonsei University Health System, Severance hospital. /ID# 141846, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 143886, Seoul
  - Samsung Medical Center /ID# 143887, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital /ID# 141844, Seoul
- Spain (7):
  - Hospital Regional de Malaga /ID# 143902, Málaga, Malaga
  - Hospital Clinic de Barcelona /ID# 143906, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 143900, Barcelona
  - Hospital Clinico Universitario San Carlos /ID# 143901, Madrid
  - Hospital Universitario 12 de Octubre /ID# 143930, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 143496, Madrid
  - Hospital General Universitario de Valencia /ID# 143903, Valencia
- Switzerland (4):
  - Kantonsspital Aarau AG /ID# 141885, Aarau, Canton of Aargau
  - Universitatsspital Zurich /ID# 141887, Zurich, Canton of Zurich
  - Duplicate_EOC Ospedale Regionale di Bellinzona e Valli /ID# 143936, Bellinzona
  - Inselspital, Universitätsspital Bern /ID# 141886, Bern
- Taiwan (3):
  - National Taiwan University Hospital /ID# 143940, Taipei
  - Taipei Veterans General Hosp /ID# 143955, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 143941, Taoyuan
- United Kingdom (9):
  - Guys and St Thomas NHS Foundation Trust /ID# 142652, London, London, City of
  - University Hospitals Birmingham NHS Foundation Trust /ID# 154592, Birmingham
  - Velindre University NHS Trust /ID# 141996, Cardiff
  - Duplicate_NHS Tayside /ID# 141651, Dundee
  - NHS Lothian /ID# 141802, Edinburgh
  - Leeds Teaching Hospitals NHS Trust /ID# 141653, Leeds
  - University College London Hospitals NHS Foundation Trust /ID# 142658, London
  - Duplicate_The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 141999, Newcastle upon Tyne
  - Royal Marsden Hospital /ID# 142827, Sutton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Lassman AB, van den Bent MJ, Gan HK, Reardon DA, Kumthekar P, Butowski N, Lwin Z, Mikkelsen T, Nabors LB, Papadopoulos KP, Penas-Prado M, Simes J, Wheeler H, Walbert T, Scott AM, Gomez E, Lee HJ, Roberts-Rapp L, Xiong H, Ansell PJ, Bain E, Holen KD, Maag D, Merrell R. Safety and efficacy of depatuxizumab mafodotin + temozolomide in patients with EGFR-amplified, recurrent glioblastoma: results from an international phase I multicenter trial. Neuro Oncol. 2019 Jan 1;21(1):106-114. doi: 10.1093/neuonc/noy091. PMID 29982805
- [Derived] Gan HK, Reardon DA, Lassman AB, Merrell R, van den Bent M, Butowski N, Lwin Z, Wheeler H, Fichtel L, Scott AM, Gomez EJ, Fischer J, Mandich H, Xiong H, Lee HJ, Munasinghe WP, Roberts-Rapp LA, Ansell PJ, Holen KD, Kumthekar P. Safety, pharmacokinetics, and antitumor response of depatuxizumab mafodotin as monotherapy or in combination with temozolomide in patients with glioblastoma. Neuro Oncol. 2018 May 18;20(6):838-847. doi: 10.1093/neuonc/nox202. PMID 29077941
- [Derived] Reardon DA, Lassman AB, van den Bent M, Kumthekar P, Merrell R, Scott AM, Fichtel L, Sulman EP, Gomez E, Fischer J, Lee HJ, Munasinghe W, Xiong H, Mandich H, Roberts-Rapp L, Ansell P, Holen KD, Gan HK. Efficacy and safety results of ABT-414 in combination with radiation and temozolomide in newly diagnosed glioblastoma. Neuro Oncol. 2017 Jul 1;19(7):965-975. doi: 10.1093/neuonc/now257. PMID 28039367
- See also: can search for the study and find research centers participating — https://www.clinicaltrialsandme.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An efficacy futility analysis, conducted in accordance with the SAP, generated a conclusive result of futility, meeting the main study's objective of determining whether the addition of Depatux-M to standard therapy improves overall survival. The study was modified at that point, remaining open until after all participants had discontinued study treatment. AbbVie therefore considered this study completed (according to the rules set out for the study) and not terminated.
Groups:
- Placebo, Radiation and Temozolomide (TMZ): Placebo is given on Day 1 of Week 1, 3 and 5 along with the standard therapy of TMZ and radiation during the chemoradiation phase. Placebo is given on Day 1 and 15 of each cycle along with TMZ (Days 1-5 of each cycle) per standard of care during the adjuvant phase.
- Depatuxizumab Mafodotin, Radiation and TMZ: Depatuxizumab mafodotin is given on Day 1 of Week 1, 3 and 5 along with the standard therapy of TMZ and radiation during the chemoradiation phase. Depatuxizumab mafodotin is given on Day 1 and 15 of each cycle along with TMZ (Days 1-5 of each cycle) per standard of care during the adjuvant phase.
Period: Overall Study
Arm/Group | Placebo, Radiation and Temozolomide (TMZ) | Depatuxizumab Mafodotin, Radiation and TMZ | Open-Label Sub-Study: Depatuxizumab Mafodotin, Radiation and TMZ
Started (Randomized) | 341 | 344 | 6
Received Randomized Study Drug | 337 | 344 | 6
Entered Adjuvant Phase | 285 | 273 | 6
Entered Follow-Up Phase | 328 | 326 | 5
Completed | 0 | 0 | 0
Not Completed | 341 | 344 | 6
Not completed — Withdrawal by Subject | 26 | 23 | 3
Not completed — Lost to Follow-up | 4 | 5 | 0
Not completed — Study Terminated by Sponsor | 107 | 89 | 2
Not completed — Death | 182 | 200 | 1
Not completed — Other, Not Specified | 20 | 27 | 0
Not completed — Unknown Reason | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Open-Label Substudy: Depatuxizumab Mafodotin, Radiation and TMZ: Depatuxizumab mafodotin is given to participants with hepatic impairment on Day 1 of Week 1, 3 and 5 along with the standard therapy of TMZ and radiation during the chemoradiation phase. Depatuxizumab mafodotin is given on Day 1 and 15 of each cycle along with TMZ (Days 1-5 of each cycle) per standard of care during the adjuvant phase.
- Total: Total of all reporting groups
Arm/Group | Placebo, Radiation and TMZ | Depatuxizumab Mafodotin, Radiation and TMZ | Open-Label Substudy: Depatuxizumab Mafodotin, Radiation and TMZ | Total
Number analyzed (Participants) | 341 | 344 | 6 | 691
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.42) | 58.2 (10.14) | 55.3 (10.58) | 58.1 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 129 | 0 | 266
  Male | 204 | 215 | 6 | 425
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 7 | 0 | 13
  Asian | 47 | 40 | 5 | 92
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 4 | 5 | 0 | 9
  White | 282 | 289 | 1 | 572
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 35 | 1 | 71
  Han Chinese (First Generation) | 28 | 23 | 2 | 53
  Other, Not Specified | 278 | 285 | 3 | 566
  Missing | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Time to OS is defined as the number of days from the date of randomization to the date of death due to any cause.
Time Frame: Overall median duration of follow-up was 15.5 months (range: 0.1, 35.6).
Population: Full Analysis Set (FAS): all randomized participants (regardless of whether they received study treatment) satisfying the following criteria:
  * Enrollment date was on or prior to 31-Mar-2018
  * Enrolled in the main study (not in the open-label hepatic sub-study)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo, Radiation and TMZ | Depatuxizumab Mafodotin, Radiation and TMZ
Number analyzed (Participants) | 316 | 323
months | 18.7 [17.0 to 20.3] | 18.9 [17.4 to 20.8]
Statistical Analysis 1: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Terms abbreviated below: O6-methylguaninemethlytransferese (MGMT); Recursive Partitioning Analysis (RPA); EGFRde2-7 (EGFRvIII); Test type: Superiority; p = 0.633, Log Rank — Weighted log-rank P-value: Stratified Fleming-Harrington (ρ = 0, γ = 0.2) test was used. Stratified by randomization stratification factors namely: MGMT methylation status, RPA class, region of the world and EGFRvIII mutation status; Cox Proportional Hazard = 1.02, 95% CI 2-sided [0.82 to 1.26] — Based on multivariate Cox proportional hazards model including treatment, MGMT methylation status, RPA class, region of the world, and EGFRvIII mutation status as covariates
Statistical Analysis 2: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Test type: Superiority; p = 0.704, Log Rank — Log-rank P-value (1-sided): Stratified by randomization stratification factors namely: MGMT methylation status, RPA class, region of the world and EGFRvIII mutation status

2. Secondary Outcome: OS for the O6-methylguaninemethlytransferese (MGMT) Unmethylated Group
Description: Time to OS is defined as the number of days from the date of randomization to the date of death due to any cause.
  Unmethylated MGMT promoter is associated with a worse prognosis in GBM
Time Frame: Overall median duration of follow-up was 15.5 months (range: 0.1, 35.6).
Population: Full Analysis Set (FAS): all randomized participants (regardless of whether they received study treatment) satisfying the following criteria:
  * Enrollment date was on or prior to 31-Mar-2018
  * Enrolled in the main study (not in the open-label hepatic sub-study) Participants with unmethylated MGMT promoter status.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo, Radiation and TMZ | Depatuxizumab Mafodotin, Radiation and TMZ
Number analyzed (Participants) | 199 | 205
months | 16.2 [14.7 to 17.7] | 16.1 [14.6 to 18.5]
Statistical Analysis 1: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Test type: Superiority; p = 0.504, Log Rank — [p-value comment as in outcome 1, analysis 1]; Cox Proportional Hazard = 0.97, 95% CI 2-sided [0.76 to 1.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Test type: Superiority; p = 0.599, Log Rank — [p-value comment as in outcome 1, analysis 2]

3. Secondary Outcome: OS for the MGMT Methylated Group
Description: Time to OS is defined as the number of days from the date of randomization to the date of death due to any cause.
Time Frame: Overall median duration of follow-up was 15.5 months (range: 0.1, 35.6).
Population: Full Analysis Set (FAS): all randomized participants (regardless of whether they received study treatment) satisfying the following criteria:
  * Enrollment date was on or prior to 31-Mar-2018
  * Enrolled in the main study (not in the open-label hepatic sub-study) Participants with methylated MGMT promoter status.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo, Radiation and TMZ | Depatuxizumab Mafodotin, Radiation and TMZ
Number analyzed (Participants) | 117 | 118
months | NA [21.2 to NA] — Median and upper limit of confidence interval not estimable due to the small number of events. | 25.4 [21.6 to 27.3]
Statistical Analysis 1: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Test type: Superiority; p = 0.773, Log Rank — [p-value comment as in outcome 1, analysis 1]; Cox Proportional Hazard = 1.17, 95% CI 2-sided [0.76 to 1.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Test type: Superiority; p = 0.740, Log Rank — [p-value comment as in outcome 1, analysis 2]

4. Secondary Outcome: OS for the Epidermal Growth Factor Receptor (EGFR)vIII-Mutated Tumor Subgroup
Description: Time to OS is defined as the number of days from the date of randomization to the date of death due to any cause.
Time Frame: Overall median duration of follow-up was 15.5 months (range: 0.1, 35.6).
Population: Full Analysis Set (FAS): all randomized participants (regardless of whether they received study treatment) satisfying the following criteria:
  * Enrollment date was on or prior to 31-Mar-2018
  * Enrolled in the main study (not in the open-label hepatic sub-study) Participants with EGFR-VIII mutation status=mutated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo, Radiation and TMZ | Depatuxizumab Mafodotin, Radiation and TMZ
Number analyzed (Participants) | 168 | 164
months | 18.2 [15.7 to 19.5] | 19.8 [17.8 to 23.1]
Statistical Analysis 1: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Test type: Superiority; p = 0.381, Log Rank — [p-value comment as in outcome 1, analysis 1]; Cox Proportional Hazard = 0.95, 95% CI 2-sided [0.71 to 1.27] — Based on multivariate Cox proportional hazards model including treatment, MGMT methylation status, RPA class, region of the world and EGFRvIII mutation status as covariates
Statistical Analysis 2: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Test type: Superiority; p = 0.409, Log Rank — [p-value comment as in outcome 1, analysis 2]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS will be defined as the number of days from the date of randomization to the date of earliest disease progression based on Response Assessment in Neuro-Oncology (RANO) criteria (see Wen et al. J Clin Oncol. 2010 Apr 10;28(11):1963-72) or to the date of death, if disease progression does not occur.
Time Frame: Overall median duration of follow-up was 15.5 months (range: 0.1, 35.6).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo, Radiation and TMZ | Depatuxizumab Mafodotin, Radiation and TMZ
Number analyzed (Participants) | 316 | 323
months | 6.3 [5.9 to 7.9] | 8.0 [6.2 to 9.6]
Statistical Analysis 1: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Test type: Superiority; p = 0.029, Log Rank — Stratified log-rank test was used. Stratified by randomization stratification factors namely: MGMT methylation status, RPA class, region of the world and EGFRvIII mutation status; Cox Proportional Hazard = 0.84, 95% CI 2-sided [0.70 to 1.01] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: PFS for EGFRvIII-Mutated Tumor Subgroup
Description: PFS will be defined as the number of days from the date of randomization to the date of earliest disease progression based on Response Assessment in Neuro-Oncology (RANO) criteria or to the date of death, if disease progression does not occur.
Time Frame: Overall median duration of follow-up was 15.5 months (range: 0.1, 35.6).
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo, Radiation and TMZ | Depatuxizumab Mafodotin, Radiation and TMZ
Number analyzed (Participants) | 168 | 164
months | 5.9 [4.8 to 7.7] | 8.3 [6.1 to 10.7]
Statistical Analysis 1: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Test type: Superiority; p = 0.002, Log Rank — [p-value comment as in outcome 5, analysis 1]; Cox Proportional Hazard = 0.72, 95% CI 2-sided [0.56 to 0.93] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Deterioration Free Survival in M.D. Anderson Symptom Inventory Brain Tumor Module (MDASI-BT) Symptom Severity Score
Description: The MDASI-BT assesses the severity of multiple brain tumor-related symptoms and the impact of these symptoms on daily functioning in the last 24 hours. It consists of 22 symptom items and 6 interference items, each rated from 0 to 10. MDASI-BT symptom severity score is defined as average over 13 core symptom items and 9 brain tumor symptom items, with a total score of 0 to 10, with higher score indicating worse symptoms/interference. Changes in symptom severity score were classified into 3 categories: improved (≤ -1), stable (> -1 and < 1), and deteriorated (≥ 1). Deterioration is defined as satisfying the deterioration criteria (i.e., increase in symptom severity score by ≥ 1 unit) without further improvement (i.e., failing to satisfy deterioration criteria) within 8 weeks or occurrence of death.
Time Frame: Overall median duration of follow-up was 15.5 months (range: 0.1, 35.6).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo, Radiation and TMZ | Depatuxizumab Mafodotin, Radiation and TMZ
Number analyzed (Participants) | 316 | 323
months | 11.0 [8.05 to 12.71] | 6.1 [4.57 to 8.02]
Statistical Analysis 1: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Test type: Superiority; p = 0.994, Log Rank — [p-value comment as in outcome 5, analysis 1]; Cox Proportional Hazard = 1.329, 95% CI 2-sided [1.087 to 1.626] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: Deterioration Free Survival in MDASI-BT Symptom Interference Score
Description: The MDASI-BT assesses the severity of multiple brain tumor-related symptoms and the impact of these symptoms on daily functioning in the last 24 hours. It consists of 22 symptom items and 6 interference items, each rated from 0 to 10. MDASI-BT symptom interference score is defined as an average of 6 interference items, with a total score of 0 to 10, where higher scores indicate worse interference. Changes in symptom interference score were classified into 3 categories: improved (≤ -1), stable (> -1 and < 1), and deteriorated (≥ 1). Deterioration is defined as satisfying the deterioration criteria (i.e., increase in symptom interference score by ≥ 1 unit) without further improvement (i.e., failing to satisfy deterioration criteria) within 8 weeks or occurrence of death.
Time Frame: Overall median duration of follow-up was 15.5 months (range: 0.1, 35.6).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo, Radiation and TMZ | Depatuxizumab Mafodotin, Radiation and TMZ
Number analyzed (Participants) | 316 | 323
months | 9.7 [7.79 to 12.19] | 6.1 [4.57 to 8.84]
Statistical Analysis 1: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Test type: Superiority; p = 0.938, Log Rank — [p-value comment as in outcome 5, analysis 1]; Cox Proportional Hazard = 1.185, 95% CI 2-sided [0.972 to 1.446] — [estimate comment as in outcome 4, analysis 1]

9. Secondary Outcome: Deterioration Free Survival in Neurocognitive Functioning on the Hopkins Verbal Learning Test Revised (HVLT-R) Total Recall Score
Description: The HVLT-R consists of 3 parts. Free call has a range of 0 to 36, delayed recall has a range from 0 to 12, and delayed recognition has a range of -12 to 12. Higher scores indicating better function in all 3 parts. When scoring the HVLT-R, the 3 learning trials are combined to calculate a total recall score (range -12 to 60). Deterioration is defined as satisfying the deterioration criteria (i.e., decrease in HVLT-R total recall score by 5 units) without further improvement within 8 weeks or occurrence of death.
Time Frame: Overall median duration of follow-up was 15.5 months (range: 0.1, 35.6).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo, Radiation and TMZ | Depatuxizumab Mafodotin, Radiation and TMZ
Number analyzed (Participants) | 316 | 323
months | 13.2 [11.53 to 14.59] | 10.7 [8.18 to 13.14]
Statistical Analysis 1: Comparison: Placebo, Radiation and TMZ vs Depatuxizumab Mafodotin, Radiation and TMZ; Test type: Superiority; p = 0.814, Log Rank — [p-value comment as in outcome 5, analysis 1]; Cox Proportional Hazard = 1.136, 95% CI 2-sided [0.921 to 1.402] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: From signing of informed consent through the end of follow-up (overall median of 17.9 months). Adverse Events: From the first dose of any study drug during each study phase and no later than 49 days after the last dose of depatuxizumab mafodotin or placebo during each study phase, or the start of a new phase. Overall, the median duration of study drug treatment was 6.0 and 7.9 months in the depatuxizumab mafodotin and placebo treatment arms, respectively.
Description: Safety Analysis Set: all randomized participants who received at least one dose of study treatment (either RT, TMZ, placebo or depatuxizumab mafodotin), classified according to treatment received. In the chemoradiation phase, 2 participants each did not have chemoradiation records in both the placebo and the depatuxizumab mafodotin arms; likewise for 2 participants in the placebo follow-up phase.
Groups:
- Placebo, Radiation and TMZ: Chemoradiation Phase: Placebo given on Day 1 of Week 1, 3 and 5 along with the standard therapy of TMZ and radiation during the chemoradiation phase.
- Placebo, Radiation and TMZ: Adjuvant Phase: Placebo given on Day 1 of Week 1, 3 and 5 along with the standard therapy of TMZ and radiation during the chemoradiation phase. Placebo given on Day 1 and 15 of each cycle, along with TMZ (Days 1-5 of each cycle) per standard of care during the adjuvant phase.
- Placebo, Radiation and TMZ: Follow Up Phase: Participants who complete placebo + TMZ adjuvant treatment or discontinue study drug prior to disease progression continue to undergo magnetic resonance imaging and assessment of neurocognitive functioning and patient reported outcomes approximately every 8 weeks up to and including at the time of disease progression, starting 8 weeks after the last scheduled assessments in the adjuvant phase. After disease progression, overall survival continues to be assessed quarterly.
- Depatuxizumab Mafodotin, Radiation and TMZ: Chemoradiation Phase: Depatuxizumab mafodotin given on Day 1 of Week 1, 3 and 5 along with the standard therapy of TMZ and radiation during the chemoradiation phase.
- Depatuxizumab Mafodotin, Radiation and TMZ: Adjuvant Phase: Depatuxizumab mafodotin given on Day 1 of Week 1, 3 and 5 along with the standard therapy of TMZ and radiation during the chemoradiation phase. Depatuxizumab mafodotin given on Day 1 and 15 of each cycle, along with TMZ (Days 1-5 of each cycle) per standard of care during the adjuvant phase.
- Depatuxizumab Mafodotin, Radiation and TMZ: Follow Up Phase: Participants who complete depatuxizumab mafodotin + TMZ adjuvant treatment or discontinue study drug prior to disease progression continue to undergo magnetic resonance imaging and assessment of neurocognitive functioning and patient reported outcomes approximately every 8 weeks up to and including at the time of disease progression, starting 8 weeks after the last scheduled assessments in the adjuvant phase. After disease progression, overall survival continues to be assessed quarterly.
- Open-Label Depatuxizumab Mafodotin, Radiation and TMZ: Chemoradiation Phase: Open-label depatuxizumab mafodotin given to participants with hepatic impairment on Day 1 of Week 1, 3 and 5 along with the standard therapy of TMZ and radiation during the chemoradiation phase.
- Open-Label Depatuxizumab Mafodotin, Radiation and TMZ: Adjuvant Phase: Open-label depatuxizumab mafodotin given to participants with hepatic impairment on Day 1 of Week 1, 3 and 5 along with the standard therapy of TMZ and radiation during the chemoradiation phase. Depatuxizumab mafodotin given on Day 1 and 15 of each cycle, along with TMZ (Days 1-5 of each cycle) per standard of care during the adjuvant phase.
- Open-Label Depatuxizumab Mafodotin, Radiation and TMZ: Follow Up Phase: Participants who complete open-label depatuxizumab mafodotin + TMZ adjuvant treatment or discontinue study drug prior to disease progression continue to undergo magnetic resonance imaging and assessment of neurocognitive functioning and patient reported outcomes approximately every 8 weeks up to and including at the time of disease progression, starting 8 weeks after the last scheduled assessments in the adjuvant phase. After disease progression, overall survival continues to be assessed quarterly.
Arm/Group | Placebo, Radiation and TMZ: Chemoradiation Phase | Placebo, Radiation and TMZ: Adjuvant Phase | Placebo, Radiation and TMZ: Follow Up Phase | Depatuxizumab Mafodotin, Radiation and TMZ: Chemoradiation Phase | Depatuxizumab Mafodotin, Radiation and TMZ: Adjuvant Phase | Depatuxizumab Mafodotin, Radiation and TMZ: Follow Up Phase | Open-Label Depatuxizumab Mafodotin, Radiation and TMZ: Chemoradiation Phase | Open-Label Depatuxizumab Mafodotin, Radiation and TMZ: Adjuvant Phase | Open-Label Depatuxizumab Mafodotin, Radiation and TMZ: Follow Up Phase
All-Cause Mortality (participants affected / at risk) | 4/335 | 13/285 | 180/326 | 4/342 | 22/273 | 188/326 | 0/6 | 0/6 | 1/5
Serious Adverse Events (participants affected / at risk) | 56/335 | 85/285 | 0/326 | 68/342 | 107/273 | 2/326 | 1/6 | 1/6 | 0/5
Other Adverse Events (participants affected / at risk) | 290/335 | 255/285 | 1/326 | 337/342 | 252/273 | 2/326 | 6/6 | 6/6 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo, Radiation and TMZ: Chemoradiation Phase (N=335) | Placebo, Radiation and TMZ: Adjuvant Phase (N=285) | Placebo, Radiation and TMZ: Follow Up Phase (N=326) | Depatuxizumab Mafodotin, Radiation and TMZ: Chemoradiation Phase (N=342) | Depatuxizumab Mafodotin, Radiation and TMZ: Adjuvant Phase (N=273) | Depatuxizumab Mafodotin, Radiation and TMZ: Follow Up Phase (N=326) | Open-Label Depatuxizumab Mafodotin, Radiation and TMZ: Chemoradiation Phase (N=6) | Open-Label Depatuxizumab Mafodotin, Radiation and TMZ: Adjuvant Phase (N=6) | Open-Label Depatuxizumab Mafodotin, Radiation and TMZ: Follow Up Phase (N=5)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APLASTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYELOSUPPRESSION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 0 (0) | 10 (14) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORNEAL DYSTROPHY (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIABETES INSIPIDUS (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATARACT NUCLEAR (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORNEAL LESION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYELID FUNCTION DISORDER (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
KERATOPATHY (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPHTHALMOPLEGIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPTIC NEUROPATHY (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ULCERATIVE KERATITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONDITION AGGRAVATED (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTHERMIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IMPAIRED HEALING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NODULAR REGENERATIVE HYPERPLASIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE HEPATITIS B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EXTRADURAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES SIMPLEX ENCEPHALITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES SIMPLEX OESOPHAGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 4 (5) | 4 (4) | 0 (0) | 3 (3) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPIDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EXPOSURE TO CONTAMINATED DEVICE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADIATION NECROSIS (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SURGICAL PROCEDURE REPEATED (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FIBRIN D DIMER INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GLOMERULAR FILTRATION RATE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOPHAGIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GLIOBLASTOMA MULTIFORME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 10 (10) | 0 (0) | 1 (1) | 9 (10) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEOPLASM SWELLING (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATAXIA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 5 (7) | 5 (5) | 0 (0) | 4 (4) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CENTRAL NERVOUS SYSTEM NECROSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL CYST (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL VENTRICLE DILATATION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CRANIAL NERVE DISORDER (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSKINESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPILEPSIA PARTIALIS CONTINUA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPILEPSY (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FACIAL PARALYSIS (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FACIAL PARESIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOCAL DYSCOGNITIVE SEIZURES (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MOTOR DYSFUNCTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROLOGICAL DECOMPENSATION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARTIAL SEIZURES (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 12 (13) | 19 (22) | 0 (0) | 11 (12) | 25 (31) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STATUS EPILEPTICUS (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VASOGENIC CEREBRAL OEDEMA (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGGRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DELIRIUM (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORGANIC BRAIN SYNDROME (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRUG REACTION WITH EOSINOPHILIA AND SYSTEMIC SYMPTOMS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EUTHANASIA (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPERFICIAL VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo, Radiation and TMZ: Chemoradiation Phase (N=335) | Placebo, Radiation and TMZ: Adjuvant Phase (N=285) | Placebo, Radiation and TMZ: Follow Up Phase (N=326) | Depatuxizumab Mafodotin, Radiation and TMZ: Chemoradiation Phase (N=342) | Depatuxizumab Mafodotin, Radiation and TMZ: Adjuvant Phase (N=273) | Depatuxizumab Mafodotin, Radiation and TMZ: Follow Up Phase (N=326) | Open-Label Depatuxizumab Mafodotin, Radiation and TMZ: Chemoradiation Phase (N=6) | Open-Label Depatuxizumab Mafodotin, Radiation and TMZ: Adjuvant Phase (N=6) | Open-Label Depatuxizumab Mafodotin, Radiation and TMZ: Follow Up Phase (N=5)
ANAEMIA (Blood and lymphatic system disorders) | 21 (29) | 14 (21) | 0 (0) | 15 (23) | 14 (27) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 21 (37) | 26 (86) | 0 (0) | 22 (35) | 22 (52) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 50 (95) | 38 (162) | 0 (0) | 36 (66) | 26 (108) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 27 (46) | 25 (49) | 0 (0) | 15 (27) | 21 (54) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 47 (80) | 75 (193) | 0 (0) | 104 (190) | 119 (343) | 0 (0) | 3 (4) | 5 (15) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 3 (3) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 3 (4) | 10 (11) | 0 (0) | 2 (2) | 13 (19) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
CORNEAL EPITHELIAL MICROCYSTS (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 22 (31) | 11 (26) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 20 (20) | 12 (12) | 0 (0) | 54 (61) | 15 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 8 (9) | 8 (9) | 0 (0) | 48 (58) | 20 (29) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
KERATITIS (Eye disorders) | 2 (2) | 3 (4) | 0 (0) | 39 (60) | 30 (91) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
KERATOPATHY (Eye disorders) | 16 (16) | 12 (17) | 0 (0) | 212 (336) | 89 (277) | 0 (0) | 6 (6) | 3 (14) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 8 (8) | 2 (2) | 0 (0) | 20 (22) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OCULAR HYPERAEMIA (Eye disorders) | 3 (3) | 2 (2) | 0 (0) | 9 (11) | 8 (12) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 16 (16) | 12 (13) | 0 (0) | 64 (89) | 33 (58) | 0 (0) | 4 (4) | 3 (8) | 0 (0)
PUNCTATE KERATITIS (Eye disorders) | 3 (3) | 7 (8) | 0 (0) | 27 (38) | 18 (50) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 21 (22) | 15 (17) | 0 (0) | 84 (97) | 38 (63) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VISUAL FIELD DEFECT (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (6) | 20 (21) | 0 (0) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 79 (89) | 51 (63) | 0 (0) | 95 (100) | 56 (65) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 16 (19) | 24 (29) | 0 (0) | 16 (18) | 21 (24) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 3 (5) | 5 (8) | 0 (0) | 5 (5) | 4 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 5 (6) | 6 (7) | 0 (0) | 7 (8) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERAESTHESIA TEETH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 79 (87) | 87 (133) | 0 (0) | 106 (130) | 64 (90) | 0 (0) | 2 (2) | 1 (3) | 0 (0)
VOMITING (Gastrointestinal disorders) | 23 (24) | 50 (63) | 0 (0) | 39 (44) | 47 (58) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 17 (22) | 17 (21) | 0 (0) | 13 (15) | 17 (21) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 8 (8) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 110 (130) | 77 (140) | 0 (0) | 132 (155) | 88 (153) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MALAISE (General disorders) | 3 (3) | 1 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 12 (12) | 12 (14) | 0 (0) | 10 (14) | 17 (19) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SWELLING (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 9 (9) | 17 (20) | 0 (0) | 5 (6) | 18 (21) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 4 (4) | 4 (5) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 7 (9) | 21 (30) | 0 (0) | 8 (9) | 19 (23) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 21 (22) | 1 (1) | 0 (0) | 18 (19) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 26 (30) | 13 (16) | 0 (0) | 57 (82) | 28 (44) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 23 (26) | 7 (7) | 0 (0) | 54 (76) | 29 (52) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 4 (4) | 0 (0) | 0 (0) | 6 (8) | 18 (27) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 7 (9) | 7 (11) | 0 (0) | 22 (39) | 45 (87) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 15 (22) | 16 (23) | 1 (1) | 12 (18) | 10 (26) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 8 (10) | 10 (17) | 0 (0) | 6 (7) | 10 (24) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 10 (12) | 14 (22) | 0 (0) | 29 (59) | 21 (47) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 7 (7) | 30 (31) | 0 (0) | 7 (7) | 27 (33) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WEIGHT INCREASED (Investigations) | 2 (3) | 8 (11) | 0 (0) | 1 (1) | 3 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 10 (20) | 17 (45) | 0 (0) | 6 (6) | 12 (21) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 36 (36) | 44 (56) | 0 (0) | 40 (44) | 42 (53) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 12 (15) | 11 (14) | 0 (0) | 9 (11) | 10 (20) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 6 (6) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (6) | 25 (32) | 0 (0) | 8 (8) | 32 (46) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 18 (18) | 0 (0) | 6 (6) | 22 (23) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 6 (7) | 9 (10) | 0 (0) | 4 (4) | 7 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 8 (9) | 12 (19) | 0 (0) | 8 (9) | 15 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 11 (12) | 0 (0) | 1 (1) | 9 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (5) | 18 (25) | 0 (0) | 4 (4) | 19 (23) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
APHASIA (Nervous system disorders) | 10 (10) | 15 (20) | 0 (0) | 7 (7) | 14 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 19 (19) | 31 (38) | 0 (0) | 11 (13) | 22 (26) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 18 (20) | 5 (5) | 0 (0) | 15 (15) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 64 (73) | 52 (80) | 0 (0) | 69 (80) | 66 (92) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 11 (13) | 21 (28) | 0 (0) | 5 (6) | 17 (25) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MEMORY IMPAIRMENT (Nervous system disorders) | 7 (7) | 21 (22) | 0 (0) | 8 (8) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 6 (7) | 17 (19) | 0 (0) | 5 (5) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAROSMIA (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 5 (5) | 5 (7) | 0 (0) | 3 (3) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 15 (16) | 19 (31) | 0 (0) | 13 (14) | 22 (42) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 5 (5) | 10 (12) | 0 (0) | 3 (4) | 14 (17) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 9 (11) | 0 (0) | 5 (5) | 18 (21) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 11 (12) | 11 (11) | 0 (0) | 11 (11) | 20 (21) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 18 (20) | 22 (25) | 0 (0) | 20 (20) | 15 (15) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 25 (26) | 0 (0) | 13 (13) | 26 (27) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 97 (103) | 10 (10) | 0 (0) | 85 (93) | 10 (11) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) | 0 (0) | 9 (9) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 17 (18) | 9 (9) | 0 (0) | 20 (20) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 14 (16) | 18 (23) | 0 (0) | 14 (15) | 21 (25) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 9 (9) | 14 (20) | 0 (0) | 16 (17) | 17 (22) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (8) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HYPERAEMIA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 8 (10) | 15 (23) | 0 (0) | 14 (15) | 18 (29) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 9 (9) | 4 (5) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-05-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT02573324/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT02573324/SAP_001.pdf